CLINICAL TRIAL: NCT04888780
Title: Gaziantep Islamic University of Science and Technology
Brief Title: Effects of Web-Based Training on HbA1c, Quality of Life and Depression Levels in Adolescents With Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gaziantep Islam Science and Technology University (Other)
Collaborators: Adiyaman University Research Hospital (Other)
Responsible Party: Principal Investigator, Sema Icel, Assistant Professor, Gaziantep Islam Science and Technology University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: GaziantepIslamicUST
Record Dates: First submitted 2021-05-07; First posted 2021-05-17 (Actual); Last update posted 2021-05-17 (Actual); Status verified 2021-05

CONDITIONS: Mental Disorder in Adolescence; Behavioral Symptoms; Problem Behavior
Keywords: Depression; Quality of life; Type 1 diabetes; Web-based training
MeSH Terms: conditions — Behavioral Symptoms; Problem Behavior; Depression; Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: The research had an experimental design with pre-test and post-test control groups. The participants were randomly assigned to the experimental and control groups.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experiment adolescent group (Experimental): The web-based Watson's Human Care Theory oriented training and support program are applied to the intervention group.
  Interventions: Other: The web-based Watson's Human Care Theory oriented training
- Control adolescent group (No Intervention): No intervention is applied to the control group.

INTERVENTIONS:
Other: The web-based Watson's Human Care Theory oriented training — Video calls were held every 15 days via the skype program with complete adherence to the schedule. In these interviews, the clinical picture of diabetes and the psychosocial status of adolescents were discussed. A total of 14 interviews with 15-day intervals were made with each adolescent. All video interviews were carried out by the first researcher and they were all recorded.
  Arms: Experiment adolescent group

SUMMARY:
Objective: This study was conducted to determine the effect of diabetes training on HbA1c, levels of depression and quality of life of Type 1 Diabetes Mellitus adolescents by using the Web-Based Watson Human Care Model.

Methods: The study was conducted with 30 adolescents between 11-18 years old who was followed by Child Endocrinology Department and who accepted to participate in the research. A web page was developed by considering Training Guide for Adolescents with Type 1 Diabetes and processes of Watson Human Care Theory. Live video interviews were done with adolescents in the experiment group on 14 sessions and these interviews were recorded.

ELIGIBILITY:
Inclusion Criteria:

* Internet access in the home environment,
* Having a computer in the home environment and being able to use a person from the child and / or family,
* Adolescent diagnosed with T1 DM at least 6 months ago,
* Adolescent's ability to understand information, read and write in Turkish, and have no problems preventing him from communicating verbally,
* Agreeing to sign the consent form that the family agreed to participate in the study,

Exclusion Criteria:

* The patients, whose families did not agree to participate in the research for various reasons,
* Internet not access in the home environment,
* Adolescent has a chronic disease other than T1 DM,
* Adolescent newly diagnosed with T1 DM,

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
Children's Depression Inventory (CDI) | 5 minutes
  CDI was developed by Kovacs in order to determine the severity of depression in children. The inventory was developed by using a language that could be easily understood by children and adolescents in ages from 6 to 17 years. It was adapted into Turkish by Öy (1990).It consists of 27 items. In each item, there are three sentences between which child or adolescent can choose by considering her/his two weeks before the application.Scores ranging from 0-2 are given to the answers given. High scores indicate the level of depression, and the highest score that can be obtained from the scale is 54. The cut-off point of the scale is 19.(Cronbach's alpha = 0.86)
Paediatric Quality of Life Inventory (PedsQL) | 5 minutes
  The Inventory was developed by Varni et al. (2003). It measures the quality of life both generally and specific to the disease. PedsQL was adapted into Turkish by Ayar and is the only type of quality of life inventory that includes scales both for the child and the parent. The inventory consists of 28 items and is divided into 5 sub-scales; which are diabetes symptoms comprising 11 items, treatment barriers comprising 4 items, treatment adherence comprising 7 items, worry comprising 3 items, and communication comprising 3 items. The high total score obtained from the scale indicates that the health-related quality of life is good. (Cronbach's alpha = 0.95)
Quality Criteria for Consumer Health Information (DISCERN) Website Evaluation Scale | 2 minutes
  DISCERN instrument; which was developed by Charnock et al. (1997) and adapted into Turkish in our country by Gokdogan and et al. (2003) was used in the research. The guide to the DISCERN quality criteria is used in order to evaluate the quality and reliability of the written materials that present health-related information. The instrument consists of 16 questions in total. The first 8 questions (1-8) in the guide evaluate the reliability of the presented information; the next 7 questions (9-15) evaluate the quality of the information about treatment and care, and the last question (16) evaluates the material in general. Each question is given a score of 1-5 (5: available, 1: unavailable).A total of 15 points indicate that the web page prepared is low in terms of information quality, and 75 points indicate high information quality.

CONTACTS AND LOCATIONS:
Locations (1):
- Adiyaman University Research Hospital, Adıyaman, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The article containing the results of the study conducted using the data of the participants is at the publishing stage.

REFERENCES:
- [Result] Karahan Okuroglu G, Ecevit Alpar S. Effect of Web-based diabetes training program on diabetes-related knowledge, attitudes, and skills of health professionals: A randomized controlled trial. Jpn J Nurs Sci. 2019 Apr;16(2):184-193. doi: 10.1111/jjns.12228. Epub 2018 Aug 2. PMID 30073784
- [Result] Jaser SS. Family interaction in pediatric diabetes. Curr Diab Rep. 2011 Dec;11(6):480-5. doi: 10.1007/s11892-011-0222-y. PMID 21853415
- [Result] Charalampopoulos D, Hesketh KR, Amin R, Paes VM, Viner RM, Stephenson T. Psycho-educational interventions for children and young people with Type 1 Diabetes in the UK: How effective are they? A systematic review and meta-analysis. PLoS One. 2017 Jun 30;12(6):e0179685. doi: 10.1371/journal.pone.0179685. eCollection 2017. PMID 28665946
- [Result] Muscatello MR, Troili GM, Pandolfo G, Mento C, Gallo G, Lanza G, Pintaudi B, Di Vieste G, Di Benedetto A, Zoccali RA, Bruno A. [Depression, anxiety and anger in patients with type 1 diabetes mellitus.]. Recenti Prog Med. 2017 Feb;108(2):77-82. doi: 10.1701/2636.27098. Italian. PMID 28287201
- [Result] McGuire HC, Ji L, Kissimova-Skarbek K, Whiting D, Aguirre F, Zhang P, Lin S, Gong C, Zhao W, Lu J, Guo X, Ji Y, Seuring T, Hong T, Chen L, Weng J, Zhou Z. Type 1 diabetes mellitus care and education in China: The 3C study of coverage, cost, and care in Beijing and Shantou. Diabetes Res Clin Pract. 2017 Jul;129:32-42. doi: 10.1016/j.diabres.2017.02.027. Epub 2017 Feb 28. PMID 28500868
- [Result] Bentzen SM, Knudsen VK, Christiensen T, Ewers B. Relative validity of a web-based food frequency questionnaire for patients with type 1 and type 2 diabetes in Denmark. Nutr Diabetes. 2016 Sep 26;6(9):e232. doi: 10.1038/nutd.2016.40. PMID 27669176
- [Result] Avdal EU, Kizilci S, Demirel N. The effects of web-based diabetes education on diabetes care results: a randomized control study. Comput Inform Nurs. 2011 Feb;29(2):101-6. doi: 10.1097/NCN.0b013e3181fcbdc6. PMID 21099675
- [Result] Knox ECL, Quirk H, Glazebrook C, Randell T, Blake H. Impact of technology-based interventions for children and young people with type 1 diabetes on key diabetes self-management behaviours and prerequisites: a systematic review. BMC Endocr Disord. 2019 Jan 10;19(1):7. doi: 10.1186/s12902-018-0331-6. PMID 30630442
- [Result] Goksen D, Atik Altinok Y, Ozen S, Demir G, Darcan S. Effects of carbohydrate counting method on metabolic control in children with type 1 diabetes mellitus. J Clin Res Pediatr Endocrinol. 2014;6(2):74-8. doi: 10.4274/Jcrpe.1191. PMID 24932599
- [Result] Bachle C, Lange K, Stahl-Pehe A, Castillo K, Holl RW, Giani G, Rosenbauer J. Associations between HbA1c and depressive symptoms in young adults with early-onset type 1 diabetes. Psychoneuroendocrinology. 2015 May;55:48-58. doi: 10.1016/j.psyneuen.2015.01.026. Epub 2015 Feb 7. PMID 25720348
- [Result] Mutlu EK, Mutlu C, Taskiran H, Ozgen IT. Association of physical activity level with depression, anxiety, and quality of life in children with type 1 diabetes mellitus. J Pediatr Endocrinol Metab. 2015 Nov 1;28(11-12):1273-8. doi: 10.1515/jpem-2015-0082. PMID 26197465
- [Result] Samardzic M, Tahirovic H, Popovic N, Popovic-Samardzic M. Health-related quality of life in children and adolescents with type 1 diabetes mellitus from Montenegro: relationship to metabolic control. J Pediatr Endocrinol Metab. 2016 Jun 1;29(6):663-8. doi: 10.1515/jpem-2015-0420. PMID 27054599
- [Result] Fredette J, Mawn B, Hood K, Fain J. Quality of Life of College Students Living With Type 1 Diabetes: A Qualitative View. West J Nurs Res. 2016 Dec;38(12):1595-1610. doi: 10.1177/0193945916651265. Epub 2016 May 25. PMID 27230752
- [Result] Demir G, Ozen S, Cetin H, Darcan S, Goksen D. Effect of Education on Impaired Hypoglycemia Awareness and Glycemic Variability in Children and Adolescents with Type 1 Diabetes Mellitus. J Clin Res Pediatr Endocrinol. 2019 May 28;11(2):189-195. doi: 10.4274/jcrpe.galenos.2019.2019.0009. Epub 2019 Jan 31. PMID 30701953
- [Result] Tektas P, Cam O. The Effects of Nursing Care Based on Watson's Theory of Human Caring on the Mental Health of Pregnant Women After a Pregnancy Loss. Arch Psychiatr Nurs. 2017 Oct;31(5):440-446. doi: 10.1016/j.apnu.2017.07.002. Epub 2017 Jul 11. No abstract available. PMID 28927506
- [Result] Arslan-Ozkan I, Okumus H, Buldukoglu K. A randomized controlled trial of the effects of nursing care based on Watson's Theory of Human Caring on distress, self-efficacy and adjustment in infertile women. J Adv Nurs. 2014 Aug;70(8):1801-12. doi: 10.1111/jan.12338. Epub 2013 Dec 22. PMID 24372443
- See also: J. Watson, Intentionality and caring-healing consciousness: a practice of transpersonal nursing. Holistic Nursing Prac. 16(4) (2002) 12-19. — https://doi.org/10.1097/00004650-200207000-00005
- See also: S.A. Fitzgerald, V.E.M. Zavala, K.Y.R. Blanco, A.P. Cupertino, M.V. Geana, E.F. Ellerbeck, Acceptability and feasibility of web-based diabetes instruction for Latinos with limited education and computer experience, JHDRP. 9(3) (2016) 94-102. — https://digitalscholarship.unlv.edu/jhdrp/vol9/iss3/6/
- See also: C. Öztürk, D. Ayar, The importance of quality of life in children with type 1 diabetes mellitus, E-Journal of Dokuz Eylul University Nursing Faculty. 6(2) (2013) 99-101. — https://dergipark.org.tr/en/pub/deuhfed/issue/46814/587063
- See also: Z. Karakus Er, Z. Özer, H. Boncuk, The effect of web based patient education on symptom management and quality of life of patients with diagnosed lung cancer. 1st International Health Sciences and Life Congress. 02-05 May, 2018. Burdur, Turkey — https://ihslc.mehmetakif.edu.tr/2018/
- See also: S. Altundağ, The effect of social support and education at adaptation to disease in children with type 1 diabetes mellitus, Pamukkale Medical Journal. 11(2) (2017) 137-144. https://doi.org/10. 5505/ptd.2017.90958. — https://dergipark.org.tr/tr/pub/patd/article/399725
- See also: E. Duras, D. Bezen, O. Özkaya, H. Dursun, Evaluation of the quality of life patients followed up with diagnosis of type 1 diabetes mellitus, The Journal of Current Pediatrics. 16(2) (2018) 72-85. — https://dergipark.org.tr/tr/pub/pediatri/issue/38632/449217
- See also: B.N.Ö. Uran, S. Ozer, Y. Yıldırım, An example of Watson's theory of human caring model: case of heart failure. Turk J Card Nur. 6(11) (2015) 183-198. https://doi.org/10.5543/khd.2015.017. — https://khd.tkd.org.tr/jvi.aspx?un=KVHD-74946
- See also: K. Öner, H. Arslantaş, Depression, internet addiction and related factors in adolescents of high school students, 6 th World Nursing and Healthcare Conference, August 15-16, 2016. London, United Kingdom.. — http://dx.doi.org/10.4172/2167-1168.C1.019